CLINICAL TRIAL: NCT02017613
Title: A Phase I, Dose Escalation Study to Evaluate Safety and Efficacy of RP6530, a Dual PI3K Delta/Gamma Inhibitor, in Patients With Relapsed or Refractory Hematologic Malignancies
Brief Title: Safety and Efficacy Study of a Dual PI3K Delta/Gamma Inhibitor in Hematological Malignancies
Acronym: PI3K
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rhizen Pharmaceuticals SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RP6530-1301; 2013-003769-32 (EudraCT Number)
Record Dates: First submitted 2013-11-26; First posted 2013-12-23 (Estimated); Last update posted 2016-06-24 (Estimated); Status verified 2016-02

CONDITIONS: Lymphoma, B-Cell; T-Cell Lymphoma
Keywords: CLL, SLL, NHL, SLL, PTCL, CTCL, MM, AML
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma, T-Cell; Lymphoma, Non-Hodgkin; Lymphoma, T-Cell, Cutaneous; Leukemia, Myeloid, Acute | interventions — tenalisib; Phosphatidylinositol 3-Kinases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single arm (Experimental): RP6530 administered orally
  Interventions: Drug: RP6530

INTERVENTIONS:
Drug: RP6530 — Escalating doses starting at 25 mg BID
  Other Names: PI3k Delta/ Gamma inhibitor

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of RP6530, a dual PI3K delta/gamma inhibitor in patients with hematologic malignancies.

DETAILED DESCRIPTION:
The Maximum tolerated dose (MTD) will be determined based on the safety, pharmacokinetic (PK) and efficacy data. Safety analyses include AE's, AE's related to the drug, SAE's, laboratory values, vitals/ ECG and dose limiting toxicity (DLT). PK include measurement of peak plasma concentration (Cmax), area under the plasma concentration versus the time curve (AUC), time of maximum concentration observed (Tmax). Efficacy analyses include overall response rate (ORR) and duration of response (DOR).

ELIGIBILITY:
Inclusion Criteria:

* Refractory to or relapsed after at least 1 prior treatment line.
* ECOG performance status ≤2
* Patients must be ≥18 years of age
* Able to give a written informed consent.

Exclusion Criteria:

* Any cancer therapy in the last 4 weeks or limited palliative radiation <2 weeks
* Patients with HBV, HCV or HIV infection
* Autologous hematologic stem cell transplant within 3 months of study entry. Allogeneic hematologic stem cell transplant within 12 months.
* Previous therapy with GS-1101 (CAL-101, idelalisib), IPI-145, TGR-1202 or any drug that specifically inhibits PI3K/ mTOR (including temsirolimus, everolimus), AKT or BTK Inhibitor (including Ibrutinib).
* Patients on immunosuppressive therapy including systemic corticosteroids.
* Patients who are receiving chronic systemic anticoagulation therapy (warfarin sodium or heparin, etc.).
* Patients with known history of liver disorders.
* Patients with uncontrolled Diabetes Type I or Type II
* Any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study.
* Women who are pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2013-11; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) and pharmacokinetics (PK) of RP6530 | 28 days
  * To access maximum tolerated dose by clinical laboratory assessments, adverse events and dose limiting toxicities.
  * PK parameter AUC, Cmax, tmax, t1/2 will be determined.

SECONDARY OUTCOMES:
Clinical response following administration of RP6530 | 8 weeks
  Overall response rate (ORR) and duration of response (DOR).

CONTACTS AND LOCATIONS:
Overall Officials: Andrés JM Ferreri, MD, Study Chair — Ospedale San Raffaele s.r.l.; Carmelo Carlo-stella, MD, Principal Investigator — Humanitas Clinical and Research Centre; Richard Delarue, MD, Principal Investigator — Hopital Necker-Enfants Malades
Locations (3):
- Rhizen Trial Site, Paris, France
- Italy (2):
  - Rhizen Trial Site 1, Milan
  - Rhizen Trial Site 2, Milan

IPD SHARING:
Plan to Share IPD: No